CLINICAL TRIAL: NCT01371422
Title: Randomized Controlled Trial Comparing the Effect of a Paravertebral Block on Pain Post Percutaneous Nephrolithotomy
Brief Title: Trial Comparing the Effect of a Paravertebral Block on Pain Post Percutaneous Nephrolithotomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was no resources to complete the study at this time
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H10-02017
Record Dates: First submitted 2011-02-10; First posted 2011-06-10 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Nephrolithiasis
Keywords: Paravertebral nerve blockade; Percutaneous nephrolithotomy/nephrolithotripsy; opioids; pain
MeSH Terms: conditions — Nephrolithiasis; Pain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (PVB) (Experimental): PVB technique will be utilized for injection of the anaesthetic under the skin before the procedure.
  Interventions: Other: Paravertebral Block (PVB)
- A2 (Placebo) (Placebo Comparator): The placebo is an inactive substance that looks identical to the test intervention but contains no active ingredients and will be administered the same as the PVB by a local skin injection, but no advancement of the needle to the paravertebral space will be made to avoid unnecessary risks.
  Interventions: Other: Saline

INTERVENTIONS:
Other: Paravertebral Block (PVB) — The T10, T11 and T12 paravertebral spaces on the operative side will be identified with ultrasound in all patients (Sonosite MicroMax, 2-5 MHz curvilinear probe).
  In the PVB group, a 90mm 22g Tuohy needle will be inserted in-plane with the live ultrasound image over the transverse process at each of these levels and 5 mL of 0.5% ropivacaine will be injected at each level.
  Arms: A1 (PVB)
Other: Saline — Ultrasonography and local infiltration of saline will only be performed
  Arms: A2 (Placebo)

SUMMARY:
This is a randomized control trial (meaning the selection is random as when flipping a coin) to assess the benefit of paravertebral blockade (PVB) in Percutaneous nephrolithotomy/nephrolithotripsy (PCNL) surgery.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy/nephrolithotripsy (PCNL) is an effective treatment that offers maximal physical removal of large kidney stones. However, despite the minimally invasive nature of the procedure, postoperative pain still remains a significant concern. General anaesthetic (solution given to put the patient to sleep) for the procedure is routinely given, along with a local anaesthetic injection at the operative site (injection of anaesthetic solution to the incision area to reduce the pain after the procedure) and pain pills to reduce the pain even further after surgery. Paravertebral nerve blockade (PVB) is a technique for inserting anesthetic solution into an area near the vertebrae (bony segments that form the spinal column of humans or backbone), and is an effective method for reducing pain in the post operative period from a variety of surgeries.

The investigators expect that the PVB can decrease side effects from opioids (pain medication) and other analgesics used post-operatively. Opioid side effects include nausea, vomiting, urinary retention, constipation, and drowsiness. Other side effects associated with anaesthetic use include peptic ulcer disease and acute renal failure. The investigators also expect that PVB will result in decreased post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* 19 or older, able to give consent
* ASA 1, 2 or 3 patients
* Patients to undergo PCNL

Exclusion Criteria:

* Complex stone with anticipation of requiring >1 access sites
* Prior diagnosis of chronic pain requiring daily opioid analgesia for > 1 month prior to diagnosis of Nephrolithiasis
* Allergy to local anesthetic
* Local infection at site of regional anesthesia
* Back or other MSK deformity that contributes to inaccuracy of paravertebral block placement
* Severe cardiopulmonary disease
* Fibromyalgia
* Anticoagulation
* Patient with language barrier or inability to communicate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours post-operative, one week post-operatively

SECONDARY OUTCOMES:
Postoperative pain measured by a visual analogue scale, length of hospital stay, and follow-up for the post operative course for complications | 1, 6, and 24 hours post-operatively
  The pain scores at each of the specific time will be compared between the PVB and no PVB arms. So we will look for differences in pain between the PVB and no-PVB group at one hour, than separately at 6 hours and than at 24 hours. Differences for each time will be looked at different time (at 1 hr than at 6 hrs than at 24 hours post-op).

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD,MSc,FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- Stone Centre, Vancouver General Hospital, Jim Pattison Pavilion, Vancouver, British Columbia, Canada